CLINICAL TRIAL: NCT04704960
Title: CirculAting Tumor DNA in Patients DIagnosed With Lung Metastasis From Colorectal Cancer: candiDate Selection for Local AblaTive thErapy
Acronym: CANDIDATE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-1176
Record Dates: First submitted 2021-01-11; First posted 2021-01-12 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Cancer; Lung Metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 20 mL of whole blood is collected and cell-free DNA is extracted
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung metastases from colorectal cancer, local ablative therapy (surgery or radiation): patients diagnosed with lung metastases from colorectal cancer and undergoing surgery or radiation for lumg metastasis
  Interventions: Other: Diagnostic Test: liquid biopsy

INTERVENTIONS:
Other: Diagnostic Test: liquid biopsy — detection of tumor DNA alteration in cf-DNA

SUMMARY:
The investigators will detect circulating tumor DNA in blood of patients with lung metastases from colorectal cancer using NGS technology and intend to use it for predicting the outcome of local treatment (surgery or radiation) and recurrence of lung metastases.

DETAILED DESCRIPTION:
The investigators produce customized gene target panel by selecting genes that are commonly found in colorectal cancer and metastasis from existing literature.

In patients diagnosed with lung metastases from colorectal cancer, 20mL of whole blood is collected before and after local treatment (surgery or radiation) and cell-free DNA (cfDNA) is extracted from the collected blood. Thereafter, 20 mL of whole blood is additionally collected once after 3 months (±2 months) and once after 6 months (±2 months) during follow-up and cfDNA is extracted. The investigators perform sequencing from the extracted cfDNA.

The investigators compare the mutations detected in cfDNA before and after local treatment and identify the trend of reducing mutations in cfDNA after local treatment. So The investigators discover biomarkers for the outcome of local treatment. The investigators also search for mutations for target drugs from mutation profiling of cfDNA.

ELIGIBILITY:
Inclusion Criteria:

1. adults over 19 years of age
2. those who understand research and have written consent
3. cases diagnosed with lung metastases from colorectal cancer

Exclusion Criteria:

1. pregnant women, nursing women
2. those who lack the ability to voluntarily agree
3. participation in other clinical trials where drugs for clinical trials are administered within the past four weeks as of the date of participation in clinical trials

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: They were diagnosed with lung metastases from colorectal cancer and are Korean. They are also treated in severance hospital during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
correlation between circulating tumor DNA (ctDNA) before and after local treatment (surgery or radiation) and recurrence of lung metastases from colorectal cancer | about 6 month but additional extension for patients with relapse after local treatment
  The investigations investigate whether ctDNA changes and f/u ctDNA fraction after local treatment (surgery or radiation) can be useful as markers to predict the outcome of local treatments.

SECONDARY OUTCOMES:
mutations related to target drug | about 6 month but additional extension for patients with relapse after local treatment
  The investigations check for target drug related mutations from mutation profiling of ctDNA.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Tae Lee, Principal Investigator — Severance Hospital
Locations (1):
- Department of Laboratory Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No